CLINICAL TRIAL: NCT05394181
Title: Notify 2: An Evaluation of the Impact of Notification of Incidental Coronary Artery Calcium on Statin Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 64798
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Notification (Experimental): Notification of the presence of at least moderate coronary artery calcium on a prior non-gated chest CT
  Interventions: Other: Notification
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Notification — Notification of patient and primary care clinician of presence of at least moderate coronary artery calcium on a prior non-gated chest CT
  Arms: Notification

SUMMARY:
The primary objective is to estimate the impact of notification of primary care provider and patient of at least moderate incidental coronary artery calcification (CAC) on a prior non-gated chest CT on statin prescription rates at 4 months among patients without a clinical history of atherosclerotic cardiovascular disease not actively on statin therapy. This study will determine if notifying patients and their primary care clinician about an existing finding will influence shared decision-making around statins between patients and their primary care clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 and less than 85
2. Non-gated chest CT from 1/1/2016-6/30/2020 with algorithm screening estimating CAC score of at least 100 Agatston Units with radiologist confirmation of moderate or severe CAC
3. Encounter with Palo Alto VA affiliated primary care since 2020

Exclusion Criteria:

1. Prior diagnosis of coronary artery disease, peripheral artery disease, or cerebrovascular disease
2. Dementia
3. Metastatic cancer or active cancer undergoing chemotherapy
4. CT coronary angiogram since 2016
5. Invasive Coronary angiogram since 2016
6. CAC scan since 2016
7. Statin therapy within prior 6 months
8. Prior ezetimibe or PCSK9 inhibitor therapy
9. Prior rhabdomyolysis with statin therapy
10. Schizophrenia
11. Substance abuse disorder (alcohol, amphetamines, cocaine, opioids)
12. Hospice
13. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Statin prescription rate | 4 months
  Prescription of statin medication

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Veteran's Affairs Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No